CLINICAL TRIAL: NCT06362733
Title: Modified Pivotal Response Treatment for Insistence on Sameness in Autistic Youth
Acronym: M-PRT-IS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Antonio Hardan, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-74165
Record Dates: First submitted 2024-03-19; First posted 2024-04-12 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder; Restricted Behavior; Autism
Keywords: Intervention; Pivotal Response Treatment
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Remote (Telehealth) Intervention Program (Experimental)
  Interventions: Behavioral: Modified Pivotal Response Treatment for Insistence on Sameness in Autistic Youth

INTERVENTIONS:
Behavioral: Modified Pivotal Response Treatment for Insistence on Sameness in Autistic Youth — This is a 12-week intervention program (1 hour/week) of treatment to target insistence on sameness in youth with autism spectrum disorder (ASD). Treatment will be delivered via secure telemedicine platform and consist of combination of parent-training and parent-mediated intervention with the child.

SUMMARY:
The purpose of this open label trial is to examine the preliminary feasibility, acceptability, and effectiveness of a 12-week behavioral intervention program (1 hour/week) to treat insistence on sameness (e.g., difficulty tolerating changes in routine) in youth with autism spectrum disorder (ASD). Treatment will be delivered via secure telemedicine platform and consist of a combination of parent-training and parent-mediated intervention with the child.

ELIGIBILITY:
Participants will include children with:

1. parent/guardian aged 18 years or older with a child aged between 4.0 to 17.11 years old at the time of parental consent;
2. diagnosed with ASD (based on history, review of available medical records including diagnostic testing, e.g., ADOS) or suspicion of ASD diagnosis and confirmed with Autism Diagnostic Interview-Revised (ADI-R);
3. parent-reported clinically significant concerns regarding insistence on sameness and behavioral inflexibility;
4. stable behavioral and pharmacological treatment for at least two weeks with no anticipated changes;
5. English-speaking parent and youth able to consistently participate in study procedures;
6. family resides in United States.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Insistence on Sameness Subscale of the Dimensional Assessment of Restricted and Repetitive Behaviors (DARB). | Screening, Baseline, every 2 weeks, 12 weeks, 24 weeks
  DARB insistence on sameness subscale scores measure insistence on sameness with higher scores indicating greater intensity of insistence on sameness. [Score Range: 0-76]

SECONDARY OUTCOMES:
Change from Baseline on Blinded Clinician Ratings of Clinical Global Impression Scale, Severity and Improvement Ratings. | Baseline, 12 weeks
  Score Range: 1 = normal, not at all ill; 7 = among the most extremely ill patients; 1 = very much informed since the initiation of treatment; 7 = very much worse since the initiation of treatment.
Change from Baseline in Parent-Rated Emotion Dysregulation on the Strengths and Difficulties Questionnaire Dysregulation Profile (SDQ-DP) during treatment. | Baseline, 6 weeks, 12 weeks, 24 weeks
  SDQ-DP indexes broad emotion dysregulation with higher scores indicating greater intensity of emotion dysregulation. [Score Range: 1-27]
Change from Baseline in Parent-Rated Behavioral Inflexibility as captured by the Behavioral Inflexibility Scale. | Baseline, 6 weeks, 12 weeks, 24 weeks
  The BIS includes 38 items with higher scores indicating greater irritability. [Score range: 0-190].
Change from Baseline in Ritualistic/Sameness Subscale of Repetitive Behavior Scale-Revised (RBS-R). | Baseline, 6 weeks, 12 weeks, 24 weeks
  Higher scores indicate higher levels of RRBs. [43 items, 12 in sameness domain]
Change from Baseline in Parent-Rated Challenging Behaviors on the Open-Source Challenging Behaviors Scale (OS-CBS). | Baseline, 12 weeks
  The OS-CBS captures the severity of categories of challenging behaviors, including property destruction, aggression, elopement, conduct problems, and self-injurious behaviors, with the option to calculate a total score for each subscale and total challenging behavior, with higher score averages indicating higher severity. [18 items]
Change from Baseline in Family Accommodation Scale - RRB (FAS-RRB). | Baseline, 6 weeks, 12 weeks
  Higher scores indicate higher levels of parental accommodation of insistence on sameness behaviors [11 items on a 5-point scale to assess frequency of accommodation behaviors].
Change from Baseline in Parent-Rated Anxiety as captured by the Anxiety Scale for Children with Autism Spectrum Disorder (ASC-ASD). | Baseline, 6 weeks, 12 weeks, 24 weeks
  ASC-ASD captures anxiety with higher scores indicating greater anxiety severity across the subdomains of separation anxiety, uncertainty, performance anxiety, and anxious arousal. [Score Range: 0-72]
Change from Baseline in Caregiver Self-Report on the Caregiver Strain Questionnaire Short Form (CGSQ-SF7). | Baseline, 12 weeks
  The CGSQ-SF7 assesses additional demands, pressures, and responsibilities in families with youths suffering from behavioral or emotional disorders, with higher scores indicating greater strain. [Score Range: 2-10]
Change from Baseline in the Caregiver Self-Report Depression, Anxiety, and Stress Scale (DASS21). | Baseline, 12 weeks
  Scores for depression, anxiety, and stress are calculated by summing the scores for the relevant items. [Scores > 34 fall in "extremely severe range']
Caregiver Report Autism Symptoms Dimension Questionnaire (ASDQ). | Baseline, Week 12
  Higher scores indicate greater levels of core autism characteristics. [Score Range: 0-39]
Caregiver Report Executive Functioning Scale (EFS). | Baseline, Week 12
  The EFS characterizes sequencing/working memory, response inhibition, set shifting, emotion regulation, and risk-taking facets of executive functioning. Higher scores indicate better executive functioning. [Score Range: 0-52]
Daily Living Skills Scale (DLSS). | Baseline, Week 12
  Higher scores indicate better ability on the DLSS. [Score Range: 0-53]

OTHER OUTCOMES:
Social Validity Measures | Week 12
  Caregivers will complete a survey and interview post-intervention to assess feasibility, acceptability, and satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hardan, MD, Principal Investigator — Stanford University
Locations (1):
- 401 Quarry Road (Remote Study), Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No